CLINICAL TRIAL: NCT04165122
Title: A Randomized, Double-Blind, Double-Dummy Phase II Study of Single Dose HDIT101 Versus Standard of Care Valaciclovir in Patients With Chronic Recurrent Anogenital HSV-2 Infection
Brief Title: Monoclonal Antibody Therapy Against Chronic Herpes Simplex Virus 2 Infection
Acronym: MATCH-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg ImmunoTherapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTX101-02G
Record Dates: First submitted 2019-11-11; First posted 2019-11-15 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Herpes Genitalis
Keywords: Herpes Genitalis
MeSH Terms: conditions — Herpes Genitalis | interventions — Valacyclovir

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Double-Dummy
Who Masked: Participant, Investigator
Masking Description: Block randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HDIT101 + Valaciclovir placebo (Experimental): Group A:
  Patients treated with a single i.v. infusion of 2 g HDIT101 for 60 min at the randomization visit and with an episodic Valaciclovir placebo bid for 3 days.
  Interventions: Biological: HDIT101; Drug: Valaciclovir placebo
- HDIT101 placebo + Valaciclovir (Active Comparator): Group B:
  Patients treated with a single i.v. infusion of HDIT101 placebo for 60 min at the randomization visit and with episodic Valaciclovir 500 mg twice daily for 3 days.
  Interventions: Drug: Valaciclovir; Biological: HDIT101 placebo

INTERVENTIONS:
Biological: HDIT101 — i.v. Infusion
  Arms: HDIT101 + Valaciclovir placebo
Drug: Valaciclovir — oral application of encapsulated Valaciclovir tablets
  Other Names: Valtrex
  Arms: HDIT101 placebo + Valaciclovir
Biological: HDIT101 placebo — i.v. Infusion
  Arms: HDIT101 placebo + Valaciclovir
Drug: Valaciclovir placebo — oral application of encapsulated Valaciclovir placebo tablets
  Arms: HDIT101 + Valaciclovir placebo

SUMMARY:
This is a randomized, double-blind, double-dummy study of single dose HDIT101 versus Standard of Care Valaciclovir.

HSV-2-positive patients with at least 4 anogenital herpes lesions in the last 12 months (or at least 2 herpes lesions with previous valaciclovir long-term therapy) can be included.

If a patients develops a anogenital Herpes lesion within 4 months after the screening visit, the patients will be randomized in a 2:1 ratio to HDIT i.v. infusion + episodic treatment with 500 mg Valaciclovir-placebo OR to a single HDIT placebo infusion + episodic treatment with 500 mg Valaciclovir orally bid for 3 days.

Study duration per patient will be 180 days starting with the randomization visit. In addition to the randomization visit, 4 visits at the site and 2 phone calls are scheduled.

At every occurence of a herpetic lesion during the study, patients are treated with Valaciclovir/ Valaciclovir-placebo and need to present at the site twice to document start and end date of the lesion (unscheduled visits).

DETAILED DESCRIPTION:
In this trial, patients with chronic recurrent herpes simplex virus (HSV-2) infections (with at least 4 herpes lesions in the last 12 months or at least 2 herpes lesions with previous valaciclovir long-term therapy) can be included.

After signature of ICF and during the screening period, the patients take daily swabs of the anogenital area for 28 days to determine HSV shedding.

Patients not developing a lesion within 4 months after screening are not randomised. Patients developing a lesion within 4 months can be randomised and the treatment must be initiated within 72 Hours upon lesion occurence.

Approximately 125 patients will be randomized in a 2:1 ratio to one of the following treatment groups:

* Arm A: single HDIT i.v. infusion applied over 1 hour at the randomization visit + episodic treatment with 500 mg Valaciclovir-placebo orally bid for 3 days.
* Arm B: single HDIT placebo i.v. infusion applied over 1 hour at the randomization visit + episodic treatment with 500 mg Valaciclovir orally bid for 3 days.

The HDIT101/HDIT101-placebo infusion is only applied once during the trial, Valaciclovir (or corresponding placebo) has to be taken upon every occurence of another Herpes lesion.

Study duration per Patient will be 180 days starting with the randomization visit. In addition to the randomization visit, 4 visits at the site and 2 phone calls are scheduled.

In case of developing another lesion after the randomization visit, patients take a single swab of the lesion and episodic SoC treatment with Valaciclovir/ Valaciclovir-placebo is started and documented in an electronic diary by the patient within 24 hours after development of first symptoms. Quality of life is also recorded.

In addition to this, the patients need to present at the site within 72 hours after occurence of a the new herpes outbreak for medical examination and to confirm the HSV-2 lesion. At this unscheduled visit at the site, the PI will take a second swab and assess the lesion (including start date). Another unscheduled visit will take place upon healing of lesion.

This procedure will be repeated for every outbreak during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing informed consent.
2. Signed informed consent for participation in the study.
3. Understanding, ability, and willingness to fully comply with study interventions and restrictions.
4. Seropositive for HSV-2.
5. History of chronic recurrent anogenital HSV-2 infection with ≥ 4 outbreaks (≥ 2 under standard suppressive antiviral therapy) in the last year with no active lesion at time of enrolment. Patients with acute lesion(s) can be enrolled when the previous lesion is healed off.
6. No use of any HSV-suppressant therapy (both approved drugs and non-approved drugs including OTC drugs) including topical applications at least 7 days prior to enrolment.
7. Willingness to not use any topical or systemic anti-HSV therapy (both approved drugs and non-approved drugs including OTC) during the study apart from the study medication.
8. Willingness to not use any topical HSV treatment upon lesion development as well as avoid any manipulation or physical impact, e.g., cooling of the lesion particularly in the prodromal stage.
9. Medical assessment with no clinically significant morbidities or abnormalities as per judgement of the investigator.
10. Women of child-bearing potential (WCBP) must have a negative beta-human chorionic gonadotropin (β-HCG) urine and/or blood test at screening and within 72 hours before receiving study treatment.
11. Willingness to use two independent effective contraceptive methods for 3 months after Visit 1. Male participants and partners of female participants have to use a condom during sexual intercourse or intimacy to reduce the probability of sexually transmitted infection.

Exclusion Criteria:

1. Patients who do not develop a lesion during the 28-day swabbing period and 3 months (90 days) afterwards (i.e., within 4 months after screening).
2. Medical history or current physical illnesses/medical conditions that constitute an unacceptable risk for study participation in the judgment of the investigator (e.g., clinically significant autoimmune disorder, active infection, uncontrolled medical conditions or organ system dysfunction that, in the investigator's opinion, could compromise the patient's safety or put the study outcomes at risk, such as uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled coronary heart disease, uncontrolled psychiatric condition).
3. Patients with herpes keratitis.
4. Immunomodulatory therapy including topical (e.g., rectal, vaginal, cutaneous, etc.) and/or oral and/or parenteral and/or inhaling steroids within 28 days before start of study treatment.
5. Any condition that precludes the sampling of up to 200 mL (additional 150 mL in case of optional participation for exploratory objective (T-cell response)) blood over the duration of the study.
6. Known resistance to or intolerance of valaciclovir or active substance or excipients of the study medication.
7. Positive HIV antibody screen, hepatitis B virus (HBV) infection screen, or hepatitis C virus (HCV) antibody screen.
8. Any known history of severe allergic or anaphylactic reactions.
9. Participation in any clinical study within the last 30 days prior to enrolment.
10. Prior participation in this or other clinical study with HDIT101.
11. Pregnant or breast-feeding women.
12. Prior malignant disease except basal cell carcinoma or carcinoma in situ which has been successfully cured more than 5 years before enrolment.
13. Hemoglobin (Hb) < 10 g/dL.
14. Creatinine (Crea) clearance (Cl) < 40 mL/min (Cockcroft-Gault equation will be used)
15. Bilirubin > upper limit of normal (ULN) x 2, except patients with known Morbus Meulengracht.
16. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > ULN x 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of days with lesion(s) per treatment group | 180 days
  Primary objective is calculated as the number of days with lesion (except the lesion episode at randomization) divided by the number of study days after IMP infusion.

SECONDARY OUTCOMES:
Time to first recurrence of lesion | 180 days
  Time to first recurrence of lesion as reported by patient and verified by investigator
Recurrence rate of lesions | 180 days
  Recurrence rate is defined as number of recurrences divided by the total number of study days after IMP infusion
Duration of recurrent lesions | 180 days
  Duration of recurrent lesions is calculated as consecutive days with lesions of HSV score 2-7
Disease-specific symptoms | 180 days
  Disease-specific symptoms assessed by Herpes Symptoms Checklist
Herpes outbreak impact | 180 days
  Herpes outbreak impact assessed by Herpes Outbreak Impact Questionnaire
QoL | 180 days
  Change in QoL between baseline and EoS assessed by the Recurrent Genital Herpes

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schoeffel, Study Director — Heidelberg ImmunoTherapeutics GmbH
Locations (8):
- Germany (8):
  - emovis GmbH, Berlin
  - Praxis Jessen2+Kollegen, Berlin
  - WIR "Walk In Ruhr" im St. Elisabeth Hospital, Bochum
  - Dr. Scholten und Schneeweiß GbR, Cologne
  - Infektio Research GmbH & Co. KG, Frankfurt
  - Universitätsklinikum Freiburg, Medizin II, Infektiologie, Freiburg im Breisgau
  - ICH Grindel, Hamburg
  - Prinzmed, München

REFERENCES:
- [Derived] Stellbrink HJ, Schaller T, Sturm K, Brockmeyer NH, Potthoff A, Bickel M, Scholten S, Postel N, Jessen A, Muller M, Jager D, Muller C, Seyfizadeh N, Schoffel S, Ullrich B, Brosi L, Kunz C, Thomas D, Laage R, Hanakam F, Schwab M, Schonborn-Kellenberger O, Mangold M, Och K, Lehr T, Arndt MA, Krauss J. Safety and efficacy of monoclonal antibody therapy in patients with chronic herpes simplex virus-2 genital infections: MATCH-2, a randomized double-blinded, parallel-group phase 2 multi-center trial. Pharmacol Res. 2025 Nov;221:107999. doi: 10.1016/j.phrs.2025.107999. Epub 2025 Oct 16. PMID 41109488